CLINICAL TRIAL: NCT06974578
Title: Assessment of the Outcomes of Routine Insertion of Capsular Tension Ring (CTR) With Hydrophilic Versus Hydrophobic Intraocular Lenses (IOLs) Alone After Phacoemulsification
Brief Title: Capsular Tension Ring With Hydeophilic Intraocular Lesnes to Decrease Posterior Capsule Opacification Versus Hydrophobic Ones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CTR with IOL
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Intraocular Lens Complication
Keywords: CTR; IOLs; Phacoemulsification
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: CTR + Hydrophilic IOL (Active Comparator): phacoemulsification and insertion of CTR the hydrophilic IOL
  Interventions: Procedure: phacoemulsification; Device: CTR; Device: hydrophilic IOL
- Group B: Hydrophobic IOL alone (Active Comparator): phacoemulsification and insertiion of hydrophobic IOL
  Interventions: Procedure: phacoemulsification; Device: Hydrophobic IOL

INTERVENTIONS:
Procedure: phacoemulsification — cataract extracton with phacoemulsification
Device: CTR — insertion of capsualr tension ring
  Arms: Group A: CTR + Hydrophilic IOL
Device: hydrophilic IOL — implantation of hydrophilic IOL
  Arms: Group A: CTR + Hydrophilic IOL
Device: Hydrophobic IOL — insertion of hydrophobic IOL
  Arms: Group B: Hydrophobic IOL alone

SUMMARY:
evaluate the clinical outcomes of routine CTR insertion in conjunction with hydrophilic versus hydrophobic IOLs following phacoemulsification.

DETAILED DESCRIPTION:
Phacoemulsification with intraocular lens (IOL) implantation is the standard surgical approach for cataract extraction. The choice between hydrophilic and hydrophobic IOLs has been debated, with studies suggesting differences in posterior capsule opacification (PCO) rates and capsular bag stability. Capsular tension rings (CTRs) are devices designed to stabilize the capsular bag, particularly in cases with zonular weakness. While CTRs are beneficial in complex cases, their routine use remains controversial. Understanding the interaction between CTRs and IOL materials could inform surgical practices and improve patient outcomes

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 40-80 years.

  * Visually significant cataract (≥3+ on Lens Opacities Classification System III "LOCSIII").
  * Clear cornea.

Exclusion Criteria:

* • Previous ocular surgery.

  * Zonular instability requiring CTR insertion beyond routine practice.
  * Complicated cataract cases (e.g., traumatic cataract).
  * Active intraocular inflammation or infection.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in BCVA (LogMAR) | at 1, 3, and 6 months postoperatively.
  The formula: logMAR score (0.1 NL + 0.02 nl) where NL = number of lines completely read and nl = number of additional letters read ap- plies. For this method, the higher the logMAR VA score, the better the visual acuity.
Refractive error measurements (spherical equivalent) | at 1, 3, and 6 months postoperatively.
  SE was calculated as the spherical power of the refractive error plus one-half of the cylinder power. Hyperopia was defined as a spherical equivalent (SE) values of ≥ + 1.00 diopter (D) and emmetropia as a SE ranging between 0.99 and - 0.49 D. Myopia was defined as a SE refraction of ≤ -0.50 D.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar Faculty of Medicine, Cairo, Egypt